CLINICAL TRIAL: NCT00250159
Title: Natural History Study of Patients With Excess Androgen
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060011; 06-CH-0011
Record Dates: First submitted 2005-11-05; First posted 2005-11-07 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-08-13

CONDITIONS: Congenital Adrenal Hyperplasia (CAH); Familial Male-Limited Precocious Puberty (FMPP)
Keywords: Congenital Adrenal Hyperplasia (CAH); Familial Male Precocious Puberty (FMPP); 21-Hydroxylase Deficiency; Adrenal Insufficiency; Natural History; Congenital Adrenal Hyperplasia; CAH; Familial Male Precocious Puberty; FMPP
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Familial Testotoxicosis; Puberty, Precocious; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1/CAH Patients Managed at the NIH: Patients with Congenital Adrenal Hyperplasia (CAH).
- 2/CAH Patients Managed by Outside Physicians: Patients with Congenital Adrenal Hyperplasia (CAH) followed by home physician post visit at NIH.
- 3/Relatives of Patients: Relatives (mostly parents) of patients will be genotyped. This is often necessary to establish the genotype of the patient.
- 4/FMPP Patients: Patients with Familial Male-Limited Precocious Puberty (FMPP).
- 5/Patients with Androgen Excess of Unknown Etiology: Patients with Androgen Excess of Unknown Etiology followed by home physician post visit at NIH.

SUMMARY:
This study will evaluate and gather information in patients with genetic causes of too much androgen (male-like hormone) in order to better understand the effects of too much androgen and describe problems associated with it. Too much androgen in childhood, if untreated, results in rapid growth and early puberty with early cessation of growth and short stature in adulthood. Too much androgen in adulthood may result in infertility, and women may have excess facial hair, acne and a more male-like appearance. Excess androgen may also affect mood and behavior and possibly the secretion of other hormones, such as insulin. Two genetic diseases that result in early childhood androgen excess are congenital adrenal hyperplasia (CAH) and familial male-limited precocious puberty (FMPP).

Patients with known or suspected CAH due to 21-hydroxylase deficiency, 11- hydroxylase deficiency, or 3-beta-hydroxysteroid dehydrogenase deficiency and males with known or suspected FMPP may be eligible for this study. Patients with both classic and non-classic CAH are eligible, and patients with androgen excess of unknown cause may be eligible.

Participants undergo the following procedures:

* Medical history and physical examination.
* Fasting blood tests for analysis of hormones, blood chemistries including blood sugar and cardiovascular risk factors such as lipids.
* Oral glucose tolerance test for patients with elevated insulin levels. For this test, a catheter (plastic tube) is placed in a vein in the patient's arm. The patient drinks a sugar-containing fluid and blood samples are collected through the catheter at intervals starting with drinking the solution, and then 30, 60 and 120 minutes after drinking the solution.
* 24-hour urine collection to measure hormone levels in the urine.
* DNA testing for patients with 21-hydroxylase deficiency to help identify the type of genetic mutation responsible for the disease.
* X-ray of the left hand to measure bone age in growing children. The x-ray is used to determine how far into puberty the child is and how much growth potential is left in the bones.
* A pelvic ultrasound in females and testicular ultrasound in males to evaluate the size and development of the gonads (ovaries in females and testes in males).
* Cognitive and psychological tests, including an IQ test and evaluation of memory, achievement and behavior.
* Other tests and evaluations based on medical need.

The schedule for these procedures varies. In a part of the study involving only patients with CAH, growing children are evaluated twice (once in childhood and once after reaching adult height), and adults are evaluated once. In another part of the study involving patients with CAH and FMPP, growing children are seen twice a year, and adults and children who have reached adult height may be seen annually. Additional visits may be scheduled if medically indicated. In this part of the study, females are asked to keep a record of their periods after their first menstrual cycle.

DETAILED DESCRIPTION:
Study Description:

Androgen excess in childhood results in pseudoprecocious puberty, accelerated childhood growth with premature epiphyseal fusion, adult short stature, and unknown metabolic and psychological perturbations. Congenital Adrenal Hyperplasia (CAH) and familial male-limited precocious puberty (FMPP) are two genetic diseases that result in early childhood androgen excess, and CAH due to 21-hydroxylase deficiency is the most common cause of hyperandrogenism in childhood. This protocol will elucidate a comprehensive phenotypic profile for patients with CAH and FMPP. Data will be collected in a large cohort of patients regarding growth and development, hormonal and metabolic factors and psychological characteristics. This protocol will allow investigators to compare patients with androgen excess of different etiologies, elucidate androgen-mediated and disease-specific phenotypic characterizations, and allow the investigators to acquire further knowledge for use in the design of future

therapeutic interventions.

Objective:

To elucidate a comprehensive phenotypic profile for patients with CAH and FMPP.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males, ages 0 - 99 with known or suspected FMPP or
  2. Patients (males and females, ages 0 - 99) with known or suspected (based on hormonal, clinical and/or genetic testing) CAH of any type.
  3. Patients with excess androgen of unknown etiology or
  4. Relatives of patients in this protocol.

EXCLUSION CRITERIA:

1. Females with isolated polycystic ovary syndrome. If, following a diagnostic work-up, a patient is determined to have PCOS as the only cause of her hyperandrogenism; she will no longer be followed on this protocol.
2. Patients with significant non-endocrine medical conditions.
3. Females who are pregnant at the time of initial enrollment.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Males, ages 0 - 99 with known or suspected FMPP
Study Population: Individuals with excess androgen, CAH, FMPP as well as their parents.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2006-01-02 (Actual)

PRIMARY OUTCOMES:
To elucidate a comprehensive phenotypic profile for patients with CAH and FMPP | Ongoing
  Better understanding of CAH and FMPP

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Merke DP, Bornstein SR. Congenital adrenal hyperplasia. Lancet. 2005 Jun 18-24;365(9477):2125-36. doi: 10.1016/S0140-6736(05)66736-0. PMID 15964450
- [Background] Grumbach MM, Shaw EB. Further studies on the treatment of congenital adrenal hyperplasia with cortisone: IV. Effect of cortisone and compound B in infants with disturbed electrolyte metabolism, by John F. Crigler Jr, MD, Samuel H. Silverman, MD, and Lawson Wilkins, MD, Pediatrics, 1952;10:397-413. Pediatrics. 1998 Jul;102(1 Pt 2):215-21. No abstract available. PMID 9651433
- [Background] Weise M, Mehlinger SL, Drinkard B, Rawson E, Charmandari E, Hiroi M, Eisenhofer G, Yanovski JA, Chrousos GP, Merke DP. Patients with classic congenital adrenal hyperplasia have decreased epinephrine reserve and defective glucose elevation in response to high-intensity exercise. J Clin Endocrinol Metab. 2004 Feb;89(2):591-7. doi: 10.1210/jc.2003-030634. PMID 14764767
- [Derived] Javaid R, Sinaii N, Kollender S, Desai J, Moon A, Merke DP. Course of COVID-19 infection in patients with congenital adrenal hyperplasia. Front Endocrinol (Lausanne). 2024 Feb 9;15:1348130. doi: 10.3389/fendo.2024.1348130. eCollection 2024. PMID 38405151
- [Derived] Lao Q, Zhou K, Parker M, Faucz FR, Merke DP. Pseudogene TNXA Variants May Interfere with the Genetic Testing of CAH-X. Genes (Basel). 2023 Jan 19;14(2):265. doi: 10.3390/genes14020265. PMID 36833192
- [Derived] Torky A, Sinaii N, Jha S, Desai J, El-Maouche D, Mallappa A, Merke DP. Cardiovascular Disease Risk Factors and Metabolic Morbidity in a Longitudinal Study of Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2021 Nov 19;106(12):e5247-e5257. doi: 10.1210/clinem/dgab133. PMID 33677504
- [Derived] Lao Q, Jardin MD, Jayakrishnan R, Ernst M, Merke DP. Complement component 4 variations may influence psychopathology risk in patients with congenital adrenal hyperplasia due to 21-hydroxylase deficiency. Hum Genet. 2018 Dec;137(11-12):955-960. doi: 10.1007/s00439-018-1959-z. Epub 2018 Nov 21. PMID 30465166
- [Derived] Turcu AF, Mallappa A, Elman MS, Avila NA, Marko J, Rao H, Tsodikov A, Auchus RJ, Merke DP. 11-Oxygenated Androgens Are Biomarkers of Adrenal Volume and Testicular Adrenal Rest Tumors in 21-Hydroxylase Deficiency. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2701-2710. doi: 10.1210/jc.2016-3989. PMID 28472487
- [Derived] Morissette R, Chen W, Perritt AF, Dreiling JL, Arai AE, Sachdev V, Hannoush H, Mallappa A, Xu Z, McDonnell NB, Quezado M, Merke DP. Broadening the Spectrum of Ehlers Danlos Syndrome in Patients With Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2015 Aug;100(8):E1143-52. doi: 10.1210/jc.2015-2232. Epub 2015 Jun 15. PMID 26075496
- [Derived] Finkielstain GP, Kim MS, Sinaii N, Nishitani M, Van Ryzin C, Hill SC, Reynolds JC, Hanna RM, Merke DP. Clinical characteristics of a cohort of 244 patients with congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2012 Dec;97(12):4429-38. doi: 10.1210/jc.2012-2102. Epub 2012 Sep 18. PMID 22990093
- [Derived] Crocker MK, Barak S, Millo CM, Beall SA, Niyyati M, Chang R, Avila NA, Van Ryzin C, Segars J, Quezado M, Merke DP. Use of PET/CT with cosyntropin stimulation to identify and localize adrenal rest tissue following adrenalectomy in a woman with congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2012 Nov;97(11):E2084-9. doi: 10.1210/jc.2012-2298. Epub 2012 Aug 17. PMID 22904181
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-CH-0011.html